CLINICAL TRIAL: NCT04308005
Title: Children's Drawing as a Measurement of Dental Anxiety in Paediatric Dentistry
Brief Title: Drawing as a Measurement of Dental Anxiety
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Collaborators: Yeditepe University (Other)
Responsible Party: Principal Investigator, ŞİRİN GÜNER ONUR, Assist. Prof. Dr., Trakya University
Other Study IDs: SONUR
Record Dates: First submitted 2019-12-25; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Dental Anxiety
Keywords: Drawing; Children; Dental Anxiety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the present study, we aimed to assess children's anxiety levels by using different dental anxiety scales and children's drawings evaluated according to two different scoring systems: Child Drawing: Hospital (CD: H) and Emotional indicators of Human Figure Drawings (HFD).

DETAILED DESCRIPTION:
Background: Drawings can be used as a method of communication that represents an individual's self-concept, anxiety, attitude, or conflict.

Aim: The purpose of this study was to evaluate children's drawing as a measure of dental anxiety in a dental setting.

Design: Seventy- eight children, aged 6-12 years, were enrolled in this study. Pulp therapy and/or restorative treatment was performed during the first therapeutic session for all participants. Sound, Eye, and Motor (SEM) and Frankl scales were used as an objective assessment of dental anxiety during treatment. After the treatment session, the children were instructed to draw a picture of a person at a dental clinic. Children's drawings were scored by a paediatric dentist and a psychologist using Child Drawing: Hospital (CD: H) scale and emotional indicators of Human Figure Drawings (HFD). The findings were compared with Frankl and SEM scores.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 years of age-independent of sex, and ethnic characteristics
* Children without previous dental treatment experience.
* Children with carious primary teeth which required pulp therapy and restorative treatment
* Children who are not considered medically compromised
* Obtained written informed consent from parents or caregivers and obtained verbal informed consent from the child for their participance in the study where procedures are explained in an age-appropriate attitude
* Children who accept to draw a picture

Exclusion Criteria:

* Children with a compromised physical and mental health history
* Children who already received dental treatments
* Children who only needed preventive treatments
* Children who reject to draw a picture

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Number of patients required was calculated on the basis of a micro-sample at an accepted level of significance(p<0.05) and a maximum permissible error α<0.05 and β<0.2. A total of 78 children were enrolled in this study. The participants of this study included children referred to, Paediatric Dentistry Department for their dental treatment on primary teeth. Once admitted to the Paediatric Dental Clinic children are examined by a paediatric dentist and each child is appointed for their dental therapeutic session. Comprehensive treatment plans of 571 children were examined and eligible 78 subjects who matched the inclusion criteria were randomly selected from children who were appointed for their first dental treatment session.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Child Drawing: Hospital (CD: H) scale | 1 hour
  Children's drawings were scored by a paediatric dentist and a psychologist using Child Drawing: Hospital (CD: H) scale.CD: H Scoring Guide, Rating Scale and the CD: H score sheet was used for the scoring of the drawings.A manual has been established to aid in scoring the drawing, which consists of specific directions and examples to assist in scoring the drawing. Raters were directed to read and understand the CD: H manual carefully, which includes the CD: H Scoring Guide and Rating Scale and the CD: H Score Sheet.The scoring of the drawing consists of three sections. Level of anxiety according to CD: H score sheet was as follows.27 <43: very low stress, 44-83: low stress, 84-129: average stress, 130-167: above average; and 168 and over: very high stress.
Human Figure Drawings (HFD) | 1 hour
  Children's drawings were scored by a paediatric dentist and a psychologist usingemotional indicators of Human Figure Drawings (HFD).Thirty clinically valid emotional indicators (EIs) consisting of 9 quality signs, 13 special features, and eight omissions.Drawings are analyzed by the presence or absence of EIs. Score EIs as 1 = present or 0 = absent, and a total score is achieved by adding all scores that can be used in statistical analysis. Drawings can be quickly evaluated for evidence of EIs which are signs on HFDs that are associated with specific traits, anxieties.For instance, insecure and anxious children prefer to draw small figures. Moreover, children with anxiety tend to shade parts of the figure.Two or more EIs imply possible emotional difficulties exhibited by the child that warrant further investigation.
Frankl Scale | 1 hour
  Frankl scale was used as an objective assessment of behaviour during treatment.The Frankl scale is rated according to the following criteria: Rating score 1: definitely negative: Refusal of treatment, crying forcefully, fearful or any other overt evidence of extreme negativism; Rating score 2: negative: Reluctant to accept treatment, uncooperative, some evidence of negative attitude but not pronounced, that is sullen, withdrawn; Rating score 3: positive: acceptance of treatment; at times cautious, willingness to comply with the dentist, at times with reservation but patient follows the dentist's direction cooperatively; Rating score 4: definitely positive: good rapport with the dentist, interested in dental procedures, laughing and enjoying the situation.
Sound, Eye, and Motor (SEM) scale | 1 hour
  Sound, Eye, and Motor (SEM) and Frankl scales were used as an objective assessment of behaviour during treatment.The slightest manifestation of the eyes, sound or motion of the patient is graded in four levels: comfort, slight discomfort, moderate pain, and pain. Rating scores range from 1 to 4. Lowest score represent comfort whereas high score indicate pain.

IPD SHARING:
Plan to Share IPD: No